CLINICAL TRIAL: NCT01303367
Title: Medication Management and Care of Demented Patients With Behavioral and Psychological Symptoms of Dementia in Taiwan: A Retrospective Pilot Study
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Winston Wu-Dien Shen, Department of Psychiatric, WanFang Hospital
Other Study IDs: 99076
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Dementia
Keywords: Dementia; behavioral and psychological symptoms of dementia
MeSH Terms: conditions — Dementia; Behavior

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- antipsychotic agents
- non-antipsychotic agents

SUMMARY:
U.S. Food and Drug Administration (FDA) and other countries issue warnings on the off-label use of antipsychotics in demented patients with behavioral and psychological symptoms of dementia (BPSD) (FDA warning, 2003; 2005; 2008). There is a significant increase in mortality rate by 1.6 fold due to cardiovascular events and aspiration pneumonia in the demented patients received antipsychotics comparing to placebo group. However, the prescription rates of antipsychotics in demented patients are still increased by 20% after several alerts in Canada (Valiyeva et al., 2008).

DETAILED DESCRIPTION:
Cumulative observations indicate that demented patients withdrawn antipsychotics may not exacerbate BPSD. The DART-AD study shows that both demented patients with/without antipsychotics for six months have no significant difference in cognitive symptoms and BPSD (Ballard et al., 2008). Moreover, the results of a long-term follow-up DART-AD study demonstrate that the survival rate of demented patients with antipsychotics is lower than those without antipsychotics at 24th month (with group vs. without group = 40% vs. 71%) and 36th month (with group vs. without group = 30% vs. 59%), respectively (Ballard et al., 2009). Recently, several studies indicate that antidepressants such as citalopram and milnacipran might be a new medication management for demented patients with BPSD (Pollock et al., 2007).

The present study is designed as a retrospective open-label pilot study. The initial research goal of this study is to determine the prevalence of psychotropic agents in demented patients in Taiwan National Health Insurance Research Database (NHIRD) (2005 v.s. 2008) and prescription rates of psychotropic agents in demented patients in Taipei Medical University-Teaching Hospitals (from 2002 to 2010). The psychotropic agents are defined as antipsychotic, antidepressant, sedative-hypnotic, anticonvulsant agents. Moreover, the second objective of this study is to investigate the risk of cardiovascular and aspiration pneumonia. Finally, the results of this study could be used to create the best and practical protocol of treatment for BPSD in demented patients of Taiwan to improve their drug safety and quality of life.

Currently, there is no treatment for BPSD, and pharmacists should recommend physicians to decrease the off-label use of antipsychotics in demented patients with BPSD. The main reason is due to the fact that off-label use of antipsychotics increases significantly the mortality rate of demented patients. The therapeutic management of BPSD should be based on the evidence-based medicine and patient safety.

ELIGIBILITY:
Inclusion Criteria:

* This study is planning to study patients with dementia (ICD-code: 290.XX), Alzheimer's disease (ICD-code: 331.0), and/or other organic psychotic conditions (chronic) (ICD-code: 294.XX), including delirium, delusion, depressive features, and/or in conditions classified elsewhere with behavior disturbance.
* This study is to include demented patients with mild to moderate cognitive impairment (mini-mental state examination [MMSE] = 10-24/ Clinical Dementia Rating [CDR] = 0.5-2).

Exclusion Criteria:

* The present proposal excludes patients with a primary history of schizophrenic disorder (ICD-code: 295XX) and bipolar disorder (296XX).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dementia patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2002-01; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winston Wu-Dien Shen, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan